CLINICAL TRIAL: NCT04158648
Title: A Multicenter, Open-Label Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Emicizumab in Patients With Mild or Moderate Hemophilia A Without FVIII Inhibitors
Brief Title: A Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Emicizumab in Participants With Mild or Moderate Hemophilia A Without FVIII Inhibitors
Acronym: HAVEN 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO41423; 2019-002179-32 (EudraCT Number); 2023-506610-52-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mild Hereditary Factor VIII Deficiency Disease Without Inhibitor; Moderate Hereditary Factor VIII Deficiency Disease Without Inhibitor; Hemophilia A
Keywords: Mild Hemophilia A Without Factor VIII Inhibitors; Moderate Hemophilia A Without Factor VIII Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emicizumab (Experimental): Participants with mild and moderate hemophilia A without factor VIII (FVIII) inhibitors will be enrolled to receive the emicizumab loading dose regimen followed by the participant's preference of one of 3 maintenance dose regimens.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Four loading doses of emicizumab 3 milligrams per kilogram of body weight (mg/kg) will be administered subcutaneously (SC) once a week (QW) for 4 weeks followed by participant's preference of one of the three following maintenance SC dose regimens: 1.5 mg/kg QW, 3 mg/kg once every 2 weeks (Q2W), or 6 mg/kg once every 4 weeks (Q4W).
  Other Names: Hemlibra; RO5534262; RG6013; ACE910

SUMMARY:
This is a multicenter, open-label, single-arm study designed to evaluate the safety, efficacy, pharmacokinetics, and pharmacodynamics of emicizumab in participants with mild or moderate hemophilia A without inhibitors against factor VIII (FVIII).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild (FVIII level between >5% and <40%) or moderate (FVIII level between ≥1% and ≤5%) congenital Hemophilia A without FVIII inhibitors
* Weight ≥3 kilograms (kg)
* Need for prophylaxis based on investigator assessment
* A negative test for inhibitor (i.e., <0.6 Bethesda Units per milliliter [BU/mL]) within 8 weeks prior to enrollment
* No documented inhibitor (i.e., <0.6 BU/mL), FVIII half-life <6 hours, or FVIII recovery <66% in the last 5 years
* Documentation of the details of prophylactic or episodic FVIII treatment and of number of bleeding episodes for at least the last 24 weeks prior to enrollment
* Adequate hematologic, hepatic, and renal function
* For women of childbearing potential: agreement to remain abstinent or use contraception (as defined in the protocol) during the treatment period and for at least 24 weeks after the final dose of study drug

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than mild or moderate congenital hemophilia A
* History of illicit drug or alcohol abuse within 48 weeks prior to screening, in the investigator's judgment
* Previous (within the last 12 months) or current treatment for thromboembolic disease or signs of thromboembolic disease
* Other conditions that may currently increase the risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Planned surgery during the emicizumab loading dose phase (surgeries in participants on emicizumab from Week 5 onwards are allowed)
* Known HIV infection with CD4 counts <200 cells per microlitre (/μL)
* Concomitant disease, condition, significant abnormality on screening evaluation or laboratory tests, or treatment that could interfere with the conduct of the study, or that would in the opinion of the investigator, pose an additional unacceptable risk in administering study drug to the participant
* Receipt of any of the following: An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration with the exception of prior emicizumab prophylaxis; A non-hemophilia-related investigational drug within last 30 days or 5 half-lives, whichever is shorter; or Any other investigational drug currently being administered or planned to be administered
* Inability to comply with the study protocol in the opinion of the investigator
* Pregnant or breastfeeding, or intending to become pregnant during the study (women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study drug)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2025-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (5):
  - Childrens Hospital LA, Los Angeles, California
  - Hemophilia of Georgia Center for Bleeding & Clotting Disorders, Atlanta, Georgia
  - Indiana Hemophilia & Thrombosis center, Indianapolis, Indiana
  - University of Michigan, C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Washington Institute for Coagulation, Seattle, Washington
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Canada (2):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Eastern Health - General Hospital, St. John's, Newfoundland and Labrador
- France (3):
  - Hopital Cardio-vasculaire Louis Pradel, Bron
  - CH de Bicetre, Le Kremlin-Bicêtre
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Germany (2):
  - Universitätsklinikum Bonn, Bonn
  - Klinikum der Universität München, Campus Innenstadt, München
- Amsterdam UMC Location AMC, Amsterdam, Netherlands
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Charlotte Maxeke Johannesburg Hospital, Johannesburg, South Africa
- Spain (2):
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (3):
  - Cardiff and Vale NHS Trust, Cardiff
  - Royal Free Hospital, London
  - Great Ormond street Hospital for Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Negrier C, Mahlangu J, Lehle M, Chowdary P, Catalani O, Bernardi RJ, Jimenez-Yuste V, Beckermann BM, Schmitt C, Ventriglia G, Windyga J, d'Oiron R, Moorehead P, Koparkar S, Teodoro V, Shapiro AD, Oldenburg J, Hermans C. Emicizumab in people with moderate or mild haemophilia A (HAVEN 6): a multicentre, open-label, single-arm, phase 3 study. Lancet Haematol. 2023 Mar;10(3):e168-e177. doi: 10.1016/S2352-3026(22)00377-5. Epub 2023 Jan 27. PMID 36716761

RESULTS

PARTICIPANT FLOW:
Groups:
- Emicizumab: Participants with mild and moderate hemophilia A without factor VIII (FVIII) inhibitors were enrolled to receive the emicizumab loading dose regimen (emicizumab 3 mg/kg administered subcutaneously [SC] QW for 4 weeks) followed by participant preference of one of the following 3 emicizumab SC maintenance dose regimens: 1.5 mg/kg QW, 3 mg/kg Q2W, or 6 mg/kg Q4W.
Period: Overall Study
Arm/Group | Emicizumab
Started (All Participants Population) | 73 (This is the number of participants who enrolled in the study.)
Received at Least One Dose of Study Drug (Treated Population) | 72 (One participant withdrew from the study prior to receiving any treatment.)
Completed 24 Weeks in the Study | 71
Completed 52 Weeks in the Study | 57
Completed | 0
Not Completed | 73
Not completed — Ongoing in the Study | 69
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The All Participants Population includes all participants who enrolled in the study.
Arm/Group | Emicizumab
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.9 (17.0)
Age, Customized [Count of Participants; unit: Participants]
  2 to <6 Years Old | 5
  6 to <12 Years Old | 11
  12 to <18 Years Old | 14
  18 to <65 Years Old | 41
  ≥65 Years Old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black or African American | 6
  White | 62
  Unknown | 2
Hemophilia A Severity [Count of Participants; unit: Participants] — Participants included in this study must have been diagnosed with mild (FVIII level between >5% and <40%) or moderate (FVIII level between ≥1% and ≤5%) congenital hemophilia A without FVIII inhibitors.
  Participants
    Mild | 21
    Moderate | 52
Emicizumab Maintenance Dosing Regimen Chosen at Enrollment [Count of Participants; unit: Participants]
  1.5 mg/kg Once Every Week (QW) | 25
  3 mg/kg Once Every 2 Weeks (Q2W) | 39
  6 mg/kg Once Every 4 Weeks (Q4W) | 8
  Not Assigned (Not Treated) | 1

OUTCOME MEASURES:

1. Primary Outcome: Model-Based Annualized Bleed Rate for Treated Bleeds
Description: The number of treated bleeds over the efficacy period was estimated as an annualized bleed rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated bleed was defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From the day of first emicizumab dose to at least 52 weeks of emicizumab treatment (median [range, min-max] efficacy period: 55.64 [8.6-89.9] weeks)
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated bleeds per year | 0.9 [0.55 to 1.52]

2. Primary Outcome: Mean Calculated Annualized Bleed Rate for Treated Bleeds
Description: The number of treated bleeds over the efficacy period is presented here as a calculated annualized bleed rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated bleed was defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated bleeds per year | 0.9 [0.02 to 5.48]

3. Primary Outcome: Median Calculated Annualized Bleed Rate for Treated Bleeds
Description: as for outcome 2
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: Treated bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated bleeds per year | 0.0 [0.00 to 0.98]

4. Secondary Outcome: Model-Based Annualized Bleed Rate for All Bleeds
Description: The number of all bleeds over the efficacy period was estimated as an annualized bleed rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule meant that two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: All bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
All bleeds per year | 2.3 [1.67 to 3.12]

5. Secondary Outcome: Mean Calculated Annualized Bleed Rate for All Bleeds
Description: The number of all bleeds over the efficacy period is presented here as a calculated annualized bleed rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule meant that two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: All bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
All bleeds per year | 2.3 [0.35 to 7.75]

6. Secondary Outcome: Median Calculated Annualized Bleed Rate for All Bleeds
Description: as for outcome 5
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: All bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
All bleeds per year | 1.0 [0.00 to 3.11]

7. Secondary Outcome: Model-Based Annualized Bleed Rate for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period was estimated as an annualized bleed rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated joint bleed was defined as a bleed with type reported as "joint" based on at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline, and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: Treated joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated joint bleeds per year | 0.2 [0.09 to 0.57]

8. Secondary Outcome: Mean Calculated Annualized Bleed Rate for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period is presented here as a calculated annualized bleed rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated joint bleed was defined as a bleed with type reported as "joint" based on at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline, and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: Treated joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated joint bleeds per year | 0.2 [0.00 to 4.15]

9. Secondary Outcome: Median Calculated Annualized Bleed Rate for Treated Joint Bleeds
Description: as for outcome 8
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: Treated joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated joint bleeds per year | 0.0 [0.00 to 0.00]

10. Secondary Outcome: Model-Based Annualized Bleed Rate for Treated Target Joint Bleeds
Description: The number of treated target joint bleeds over the efficacy period was estimated as an annualized bleed rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated target joint bleed was defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry or an unresolved target joint (target joint that does not fulfil ≤2 bleeds into this joint within a consecutive 12-month period), and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: Treated target joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated target joint bleeds per year | 0.1 [0.03 to 0.40]

11. Secondary Outcome: Mean Calculated Annualized Bleed Rate for Treated Target Joint Bleeds
Description: The number of treated target joint bleeds over the efficacy period is presented here as a calculated annualized bleed rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated target joint bleed was defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry or an unresolved target joint (target joint that does not fulfil ≤2 bleeds into this joint within a consecutive 12-month period), and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: Treated target joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated target joint bleeds per year | 0.1 [0.00 to 3.92]

12. Secondary Outcome: Median Calculated Annualized Bleed Rate for Treated Target Joint Bleeds
Description: as for outcome 11
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: Treated target joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated target joint bleeds per year | 0.0 [0.00 to 0.00]

13. Secondary Outcome: Model-Based Annualized Bleed Rate for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period was estimated as an annualized bleed rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated spontaneous bleed was defined as a treated bleed (bleed directly followed by a hemophilia medication reported to be a "treatment for bleed") with no other known contributing factor such as trauma or procedure/surgery. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: Treated spontaneous bleeds
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated spontaneous bleeds | 0.2 [0.11 to 0.33]

14. Secondary Outcome: Mean Calculated Annualized Bleed Rate for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period is presented here as a calculated annualized bleed rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated spontaneous bleed was defined as a treated bleed (bleed directly followed by a hemophilia medication reported to be a "treatment for bleed") with no other known contributing factor such as trauma or procedure/surgery. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: Treated spontaneous bleeds
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated spontaneous bleeds | 0.3 [0.00 to 4.23]

15. Secondary Outcome: Median Calculated Annualized Bleed Rate for Treated Spontaneous Bleeds
Description: as for outcome 14
Time Frame: as for outcome 1
Population: The Treated Population comprises all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: Treated spontaneous bleeds
Arm/Group | Emicizumab
Number analyzed (Participants) | 72
Treated spontaneous bleeds | 0.0 [0.00 to 0.00]

16. Secondary Outcome: CATCH Questionnaire for Adult Participants: Change From Baseline in the Daily Activity Risk Perception and Impact Domain Scores Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: Baseline (Week 1), Weeks 13, 25, 37 and 49, and every 12 weeks thereafter until Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

17. Secondary Outcome: CATCH Questionnaire for Adult Participants: Change From Baseline in the Social Activity Risk Perception and Impact Domain Scores Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

18. Secondary Outcome: CATCH Questionnaire for Adult Participants: Change From Baseline in the Recreational Activity Risk Perception and Impact Domain Scores Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

19. Secondary Outcome: CATCH Questionnaire for Adult Participants: Change From Baseline in the Work Impact Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

20. Secondary Outcome: CATCH Questionnaire for Adult Participants: Change From Baseline in the Preoccupation Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

21. Secondary Outcome: CATCH Questionnaire for Adult Participants: Change From Baseline in the Treatment Burden Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

22. Secondary Outcome: CATCH Questionnaire for Adult Participants: Number of Participants by Responses to Their Level of Pain Associated With a Bleed Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

23. Secondary Outcome: CATCH Questionnaire for Adult Participants: Number of Participants by Responses to Their Level of Pain in Target Joints Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

24. Secondary Outcome: CATCH Questionnaire for Adult Participants: Number of Participants by Responses to Their Level of Pain at Its Worst Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

25. Secondary Outcome: CATCH Questionnaire for Adult Participants: Number of Participants by Responses to Their Level of Pain at Its Least Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

26. Secondary Outcome: CATCH Questionnaire for Adult Participants: Number of Participants by Responses to Their Level of Pain on Average Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

27. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Change From Baseline in the Daily Activity Risk Perception and Impact Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

28. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Change From Baseline in the Social Activity Risk Perception and Impact Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

29. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Change From Baseline in the Recreational Activity Risk Perception and Impact Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

30. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Change From Baseline in the School Impact Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

31. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Change From Baseline in the Preoccupation Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

32. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Change From Baseline in the Treatment Burden Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

33. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Number of Participants by Responses to Their Level of Pain Associated With a Bleed Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

34. Secondary Outcome: CATCH Questionnaire for Pediatric Participants: Number of Participants by Responses to Their Level of Pain at Its Worst Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

35. Secondary Outcome: CATCH Questionnaire for Caregivers: Change From Baseline in the Preoccupation Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

36. Secondary Outcome: CATCH Questionnaire for Caregivers: Change From Baseline in the Treatment Burden Domain Score Over Time
Description: CATCH = Comprehensive Assessment Tool of Challenges in Hemophilia
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-12

37. Secondary Outcome: Percentage of Participants Who Prefer Emicizumab SC Treatment, Their Previous Hemophilia IV Treatment, or Have No Preference, as Assessed Through Use of the Emicizumab Preference Survey at Week 17
Description: The Emicizumab Preference Survey is a fit-for-purpose questionnaire developed by the sponsor to record the participant's preference for treatment with subcutaneous (SC) emicizumab, intravenous (IV) factor VIIII (FVIII), or no preference. The 95% confidence intervals were calculated using the Pearson-Clopper method.
Time Frame: Week 17
Population: The analysis population included all treated participants 12 years of age or older who provided a response to the survey at Week 17.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 52
Percentage of participants
  Prefer the New Study Drug Treatment (Emicizumab SC) | 96.2 [86.79 to 99.53]
  Prefer My Old Hemophilia Treatment (IV) | 1.9 [0.05 to 10.26]
  Have No Preference | 1.9 [0.05 to 10.26]

38. Secondary Outcome: Percentage of Caregivers Who Prefer Emicizumab SC Treatment, Their Child's Previous Hemophilia IV Treatment, or Have No Preference, as Assessed Through Use of the Emicizumab Preference Survey at Week 17
Description: The Emicizumab Preference Survey is a fit-for-purpose questionnaire developed by the sponsor to record the caregiver's preference for their child's treatment with subcutaneous (SC) emicizumab, intravenous (IV) factor VIIII (FVIII), or no preference. The 95% confidence intervals were calculated using the Pearson-Clopper method.
Time Frame: Week 17
Population: The analysis population included all caregivers of treated participants less than 18 years of age and who provided a response to the survey at Week 17.
Measure: Number (95% Confidence Interval); unit: Percentage of caregivers
Arm/Group | Emicizumab
Number analyzed (Participants) | 28
Percentage of caregivers
  Prefer the New Study Drug Treatment (Emicizumab SC) | 85.7 [67.33 to 95.97]
  Prefer My Child's Old Hemophilia Treatment (IV) | 3.6 [0.09 to 18.35]
  Have No Preference | 10.7 [2.27 to 28.23]

39. Secondary Outcome: Hemophilia Joint Health Scores Over Time
Time Frame: Days -7 to -1, Weeks 25, 49, and every 24 weeks thereafter until Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

40. Secondary Outcome: Change From Baseline in Mean Daily Peak Activity Duration Over Time
Description: For physical activity assessment, participants ≥5 years of age were instructed to wear the study accelerometry device on the wrist continuously (24 hours/day) every day for the designated 2-week periods during the study. A participant was considered to be compliant with the physical activity assessments if they wore the study device continuously (≥8 hours/day) every day for at least 8 days of each of the designated 2-week periods during the study. If this compliance criterion was not reached at a specific timepoint the participant was not included in the analysis of the designated 2-week periods where compliance was not reached. Daily measurements were averaged over the 14-days timepoint. Activity count was a measure of the acceleration measured by the device. The daily peak activity duration was defined as the sum of moderate to vigorous activity per day (in minutes).
Time Frame: Baseline (Weeks 1-2) and Weeks 13 (Weeks 12-13 period), 25 (Weeks 24-25 period), 37 (Weeks 36-37 period), and 49 (Weeks 48-49 period)
Population: The analysis population is treated participants ≥5 years old, further subdivided into analysis groups of ≥5 to <18 years old and ≥18 years old. The number analyzed for change from baseline (BL) are participants with data that met the compliance criterion at BL and the specified timepoint (i.e., wearing device ≥8 hours/day for ≥8 days per period); if it was not met, they were excluded for each noncompliant timepoint. The overall number analyzed had valid data for at least the BL timepoint.
Measure: Mean (Standard Deviation); unit: Minutes per day
Groups:
- Participants ≥5 Years Old: Emicizumab; Participants ≥5 to <18 Years Old: Emicizumab; Participants ≥18 Years Old: Emicizumab: Participants with mild and moderate hemophilia A without factor VIII (FVIII) inhibitors were enrolled and received the emicizumab loading dose regimen (emicizumab 3 mg/kg administered subcutaneously QW for 4 weeks) followed by participant preference of one of the following 3 emicizumab maintenance dose regimens: 1.5 mg/kg QW, 3 mg/kg Q2W, or 6 mg/kg Q4W.
Arm/Group | Participants ≥5 Years Old: Emicizumab | Participants ≥5 to <18 Years Old: Emicizumab | Participants ≥18 Years Old: Emicizumab
Number analyzed (Participants) | 61 | 22 | 39
Minutes per day
  Baseline (BL) - Value at Visit | 130 (56) | 168 (66) | 108 (35)
  Change from BL at Week 13: number analyzed (Participants) | 51 | 21 | 30
  Change from BL at Week 13 | -2 (34) | -4 (42) | -1 (29)
  Change from BL at Week 25: number analyzed (Participants) | 50 | 18 | 32
  Change from BL at Week 25 | 4 (53) | -4 (74) | 8 (37)
  Change from BL at Week 37: number analyzed (Participants) | 51 | 20 | 31
  Change from BL at Week 37 | 14 (55) | 17 (73) | 12 (40)
  Change from BL at Week 49: number analyzed (Participants) | 47 | 17 | 30
  Change from BL at Week 49 | 17 (40) | 19 (51) | 16 (34)

41. Secondary Outcome: Change From Baseline in Mean Daily Step Count Over Time
Description: For physical activity assessment, participants ≥5 years of age were instructed to wear the study accelerometry device on the wrist continuously (24 hours/day) every day for the designated 2-week periods during the study. A participant was considered to be compliant with the physical activity assessments if they wore the study device continuously (≥8 hours/day) every day for at least 8 days of each of the designated 2-week periods during the study. If this compliance criterion was not reached at a specific timepoint the participant was not included in the analysis of the designated 2-week periods where compliance was not reached. Daily measurements were averaged over the 14-days timepoint. Activity count was a measure of the acceleration measured by the device.
Time Frame: Baseline (Weeks 1-2) and Weeks 13 (Weeks 12-13), 25 (Weeks 24-25), 37 (Weeks 36-37), and 49 (Weeks 48-49)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Step count per day
Arm/Group | Participants ≥5 Years Old: Emicizumab | Participants ≥5 to <18 Years Old: Emicizumab | Participants ≥18 Years Old: Emicizumab
Number analyzed (Participants) | 61 | 22 | 39
Step count per day
  Baseline (BL) - Value at Visit | 6441 (2617) | 6755 (3168) | 6263 (2276)
  Change from BL at Week 13: number analyzed (Participants) | 51 | 21 | 30
  Change from BL at Week 13 | 44 (1846) | -18 (2361) | 87 (1423)
  Change from BL at Week 25: number analyzed (Participants) | 50 | 18 | 32
  Change from BL at Week 25 | 119 (2977) | -69 (4348) | 225 (1901)
  Change from BL at Week 37: number analyzed (Participants) | 51 | 20 | 31
  Change from BL at Week 37 | 767 (3189) | 1403 (4544) | 356 (1852)
  Change from BL at Week 49: number analyzed (Participants) | 47 | 17 | 30
  Change from BL at Week 49 | 1216 (2440) | 1740 (3130) | 919 (1945)

42. Secondary Outcome: Menstrual Bleed Questionnaire (MBQ) for Female Participants of Childbearing Potential: Change From Baseline in the MBQ Total Score Over Time
Time Frame: Baseline (Week 1), Weeks 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and every 4 weeks thereafter until Study Completion (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

43. Secondary Outcome: Menstrual Bleed Questionnaire (MBQ) for Female Participants of Childbearing Potential: Change From Baseline in the Heaviness Subscale Score Over Time
Time Frame: as for outcome 42
Reporting Status: Not Posted, anticipated posting 2026-12

44. Secondary Outcome: Menstrual Bleed Questionnaire (MBQ) for Female Participants of Childbearing Potential: Change From Baseline in the Quality of Life Subscale Score Over Time
Time Frame: as for outcome 42
Reporting Status: Not Posted, anticipated posting 2026-12

45. Secondary Outcome: Menstrual Bleed Questionnaire (MBQ) for Female Participants of Childbearing Potential: Change From Baseline in the Irregularity Subscale Score Over Time
Time Frame: as for outcome 42
Reporting Status: Not Posted, anticipated posting 2026-12

46. Secondary Outcome: Menstrual Bleed Questionnaire (MBQ) for Female Participants of Childbearing Potential: Change From Baseline in the Pain Subscale Score Over Time
Time Frame: as for outcome 42
Reporting Status: Not Posted, anticipated posting 2026-12

47. Secondary Outcome: Menstruation Diary With the Pictorial Blood Assessment Chart (PBAC) for Female Participants of Childbearing Potential: PBAC Scores Over Time
Time Frame: Baseline (Day 1) and monthly (on days of menstruation) until Study Completion (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

48. Secondary Outcome: Number of Participants With at Least One Adverse Event by Severity, According to the World Health Organization (WHO) Toxicity Grading Scale
Time Frame: From Screening (Day -28 to -1) to Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

49. Secondary Outcome: Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Time Frame: From Screening (Day -28 to -1) to Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

50. Secondary Outcome: Number of Participants With at Least One Thromboembolic Event
Time Frame: From Screening (Day -28 to -1) to Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

51. Secondary Outcome: Number of Participants With at Least One Event of Thrombotic Microangiopathy
Time Frame: From Screening (Day -28 to -1) to Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

52. Secondary Outcome: Number of Participants With at Least One Injection-Site Reaction by Severity, According to the WHO Toxicity Grading Scale
Time Frame: From Screening (Day -28 to -1) to Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

53. Secondary Outcome: Number of Participants With at Least One Severe Hypersensitivity, Anaphylaxis, and Anaphylactoid Event
Time Frame: From Screening (Day -28 to -1) to Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

54. Secondary Outcome: Number of Participants With at Least One Laboratory Abnormality
Description: Laboratory parameters for hematology and blood chemistry will be measured and compared with a standard reference range. Values outside the standard reference range are considered abnormalities. Not every laboratory abnormality qualifies as an adverse event. A laboratory test result will be reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment or a medical intervention; or is clinically significant in the investigator's judgment.
Time Frame: From Screening (Day -28 to -1) to Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

55. Secondary Outcome: Change From Baseline in Respiratory Rate Over Time
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, and 49, and every 12 weeks thereafter until Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

56. Secondary Outcome: Change From Baseline in Pulse Rate Over Time
Time Frame: as for outcome 55
Reporting Status: Not Posted, anticipated posting 2026-12

57. Secondary Outcome: Change From Baseline in Body Temperature Over Time
Time Frame: as for outcome 55
Reporting Status: Not Posted, anticipated posting 2026-12

58. Secondary Outcome: Change From Baseline in Systolic Blood Pressure Over Time
Time Frame: as for outcome 55
Reporting Status: Not Posted, anticipated posting 2026-12

59. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure Over Time
Time Frame: as for outcome 55
Reporting Status: Not Posted, anticipated posting 2026-12

60. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters Over Time: QT, QTcB, QTcF, RR, PR, and QRS Intervals
Time Frame: Baseline, Weeks 5, 25, and 49, and every 12 weeks thereafter until Study Completion/Discontinuation Visit (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

61. Secondary Outcome: Change From Baseline in Heart Rate Over Time, as Measured by Electrocardiogram (ECG)
Time Frame: as for outcome 60
Reporting Status: Not Posted, anticipated posting 2026-12

62. Secondary Outcome: Plasma Trough Concentration (Ctrough) of Emicizumab Over Time
Time Frame: Pre-dose at Weeks 1, 2, 3, 4, 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, and 49, and every 12 weeks thereafter until study completion/discontinuation (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

63. Secondary Outcome: Number of Participants With Anti-Drug Antibodies Against Emicizumab at Baseline and Post-Baseline
Time Frame: Pre-dose at Baseline (Week 1) and Weeks 5, 13, 25, 33, 41, and 49, and every 12 weeks thereafter until study completion/discontinuation (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

64. Secondary Outcome: Number of Participants Who Develop Anti-FVIII Inhibitors Over Time
Time Frame: Screening (Day -28 to -1) and Weeks 1, 13, 25, 37, and 49, and every 12 weeks thereafter until study completion/discontinuation (up to approximately 48 months)
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: From enrollment until primary completion date cutoff (median [range, min-max] observation period: 55.64 [8.7-89.9] weeks)
Description: Adverse events (AEs) are reported in the Treated Population, comprising all participants who received at least one dose of emicizumab. AEs are still being collected until the end of the study and the results will be updated within 1 year of the date of final data collection.
Arm/Group | Emicizumab
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 8/72
Other Adverse Events (participants affected / at risk) | 37/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emicizumab (N=72)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emicizumab (N=72)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Injection site reaction (General disorders) | 12 (29)
Headache (Nervous system disorders) | 12 (16)
COVID-19 (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 5 (8)
Fall (Injury, poisoning and procedural complications) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT04158648/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT04158648/SAP_001.pdf